CLINICAL TRIAL: NCT07255638
Title: A Prospective Non-Interventional Study to Describe the Effectiveness of Avapritinib (BLU-285), a Selective KIT Mutation-Targeted Tyrosine Kinase Inhibitor, in Patients With Indolent Systemic Mastocytosis and Symptoms That Are Not Adequately Controlled With Symptomatic Treatments in Real-World Settings
Brief Title: A Non-Interventional Study in Participants With Indolent Systemic Mastocytosis (ISM) in Germany
Status: Recruiting | Type: Observational
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BLU-285-2407
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Indolent Systemic Mastocytosis
Keywords: ISM; Indolent systemic mastocytosis; Avapritinib; BLU-285; Selective KIT mutation-targeted tyrosine kinase inhibitor; Tyrosine kinase inhibitor; Mastocytosis; Neoplastic mast cells
MeSH Terms: conditions — Mastocytosis, Systemic; Mastocytosis | interventions — avapritinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Avapritinib: Participants will receive avapritinib as part of their treatment plan with their healthcare practitioner (HCP) and in accordance with the Summary of Product Characteristics (SmPC).
  Interventions: Drug: Avapritinib

INTERVENTIONS:
Drug: Avapritinib — Avapritinib will be administered as an oral tablet.
  Other Names: Ayvakyt; BLU-285

SUMMARY:
This is a non-interventional study assessing the effectiveness of avapritinib (BLU-285) in the management of ISM in real-world settings in Germany. The study also seeks to address the existing data gap in the natural history and management of participants with ISM.

The study is designed to follow each participant up to a maximum of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants is starting avapritinib treatment at the HCP's discretion as part of their routine care (for ISM with moderate to severe symptoms inadequately controlled with symptomatic treatment) and in accordance with approved SmPC.

Exclusion Criteria:

* Participant with a potential increased risk for intracranial hemorrhage including those with a history of vascular aneurysm, intracranial hemorrhage, cerebrovascular accident within the prior year, or severe thrombocytopenia.
* Participant who has previously taken avapritinib as a commercial drug or as part of a clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with ISM with moderate to severe symptoms inadequately controlled on symptomatic treatment, who are initiating treatment with commercial avapritinib according to the German approved label.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Mastocytosis Control-quality of Life (MC-QoL) Questionnaire Score at Month 6 | Baseline, Month 6

SECONDARY OUTCOMES:
Socio-demographic Variable: Participant Age | Baseline (Day -30 to Day -1)
Socio-demographic Variable: Participant Gender | Baseline (Day -30 to Day -1)
Socio-demographic Variable: Participant Ethnicity | Baseline (Day -30 to Day -1)
Socio-demographic Variable: Participant Race | Baseline (Day -30 to Day -1)
Baseline Serum Tryptase and KIT D816V Variant Allele Fraction (VAF) | Baseline (Day -30 to Day -1)
Number of Participants With Prior Medical History of Anaphylaxis | Baseline (Day -30 to Day -1)
Number of Participants with Comorbidity | Baseline up to Month 24
Number of Participants Initiating a New ISM-directed Medication, Discontinuing an ISM-directed Medication, and With Dose Increases or Decreases for ISM-directed Medications | Baseline up to Month 24
Number of Participants Prescribed a Life Support Kit | Baseline up to Month 24
Change From Baseline in Mastocytosis Activity Score (MAS) at Months 3, 6, 12, 18, and 24 | Baseline, Months 3, 6, 12, 18, and 24
Change From Baseline in MC-QoL Questionnaire Score at Months 3, 6, 12, 18, and 24 | Baseline, Months 3, 6, 12, 18, and 24
Change From Baseline in Mastocytosis Control Test (MCT) Score at Months 3, 6, 12, 18, and 24 | Baseline, Months 3, 6, 12, 18, and 24
Time to Response as Assessed by MAS | Baseline up to Month 24
Change From Baseline in Serum Tryptase at Months 3, 6, 12, 18, and 24 | Baseline, Months 3, 6, 12, 18, and 24
Number of Participants With Anaphylaxis Requiring Hospitalization, Emergency Room (ER) Visit, Epinephrine Autoinjector Use, or Other Medication | Baseline up to Month 24
Number of Participants Meeting the Definition of Polypharmacy (Use of Multiple Medications Simultaneously; Typically, 3 or More Symptom-directed Prescription Drugs) | Baseline up to Month 24
Number of Participants With ISM-related Hospital Visits and ER Visits | Baseline up to Month 24
Number of Participants With Changes in ISM Symptom-directed Therapies | Baseline up to Month 24
Number of Participants With Dose Modifications and Study/Treatment Discontinuations | Baseline up to Month 24

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Charité Universitätmedizin Berlin, Klinik für Dermatologie, Venerologie und Allergologie, Berlin
  - Universitätsklinikum Carl Gustav Carus Dresden Klinik und Poliklinik für Dermatologie, Dresden
  - University Medical Center Goettingen - Georg August University of Goettingen, Göttingen
  - Universitats-Hautklinik Tubingen, Studienzentrum lmmundermatologie, Tübingen